CLINICAL TRIAL: NCT03168568
Title: Differential Vascular and Endocrine Effects of Valsartan/Sacubitril in Heart Failure With Reduced Ejection Fraction: A Double-blind Randomized Controlled Phase IV Trial (VASCEND)
Brief Title: Differential Vascular and Endocrine Effects of Valsartan/Sacubitril in Heart Failure With Reduced Ejection Fraction
Acronym: VASCEND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VASCEND
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Valsartan; sacubitril; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsartan/Sacubitril (Experimental): Valsartan-Sacubitril 50mg/100mg twice daily, titrated to 200mg twice daily p.o. Duration of product administration: 3 months
  Interventions: Drug: Valsartan/Sacubitril or placebo
- Valsartan (Active Comparator): Valsartan 40mg/80mg twice daily, titrated to 160mg twice daily p.o Duration of product administration: 3 months
  Interventions: Drug: Valsartan or placebo

INTERVENTIONS:
Drug: Valsartan/Sacubitril or placebo — tablet (double dummy)
  Other Names: Entresto®; LCZ696
  Arms: Valsartan/Sacubitril
Drug: Valsartan or placebo — tablet (double dummy)
  Other Names: Diovan®
  Arms: Valsartan

SUMMARY:
The objective of this study is to evaluate whether valsartan/sacubitril leads to a superior improvement in endothelial function and endocrine status compared to valsartan alone.

DETAILED DESCRIPTION:
Valsartan/sacubitril (Entresto®; LCZ696) is a first-in-class angiotensin receptor neprilysin inhibitor (ARNI) that has recently been approved for the treatment of chronic heart failure with reduced ejection fraction (HFrEF). The drug consists of a 1:1 complex of the angiotensin receptor blocker (ARB) valsartan and the neprilysin inhibitor sacubitril. In a recent randomized controlled trial in patients with heart failure and reduced ejection fraction (PARADIGM-HF), valsartan/sacubitril significantly reduced all-cause and cardiovascular mortality as well as hospitalizations for heart failure compared to enalapril. The precise reason why combined angiotensin receptor and neprilysin blockade is superior to ACE blockade is still unclear and knowledge of the mechanisms involved would provide further insight which patients with symptomatic heart failure will particularly benefit from valsartan/sacubitril. On the one hand, many of the peptides affected by neprilysin blockade act on vascular endothelial cells. On the other, neprilysin inhibition may induce significant endocrine changes with a shift to more favorable hormonal profile in HFrEF patients. Detailed studies on the vascular and endocrine effects of valsartan/sacubitril in humans are lacking so far. The investigators hypothesize that valsartan/sacubitril results in an incremental improvement of endothelial dysfunction and endocrine imbalance over valsartan in patients with heart failure with reduced ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age, male or female, with a diagnosis of symptomatic heart failure (NYHA class II-IV) per ESC heart failure guidelines
2. LVEF ≤ 40%
3. Established guideline-recommended therapy with an ACEI, ARB and a beta-blocker, as clinically indicated and tolerated, at stable doses for at least 3 weeks prior to inclusion.

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the study drugs
2. History of angioedema.
3. Sitting systolic blood pressure <90 mmHg at Visit 1 (screening) or Visit 2 (randomization)
4. Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy).
5. Estimated GFR < 20 mL/min/1.73m2
6. Serum potassium > 5.5 mmol/L at Visit 1 (screening) or Visit 2 (randomization).
7. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major CV surgery, percutaneous coronary intervention (PCI) or carotid angioplasty within the 3 months prior to Visit 1.
8. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 3 months after Visit 1.
9. Implantation of a cardiac resynchronization therapy device (CRTD) within 2 months prior Visit 1 or intent to implant a CRTD within next 3 months.
10. History of heart transplant, on a transplant list or with ventricular assistance device (VAD).
11. Presence of significant endocrine diseases.
12. Presence of active acute infectious diseases.
13. Known narrow-angle glaucoma
14. Known epilepsy
15. Cimino-shunt operation on both arms
16. Pregnancy, intention thereof during study; lack of sufficient contraception; breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Difference in flow-mediated vasodilatation (FMD) | Baseline, 3 months
  Difference in flow-mediated vasodilatation (FMD, percent dilatation of brachial artery after blood pressure cuff occlusion) between the valsartan/sacubitril and valsartan group as assessed at the final study visit

SECONDARY OUTCOMES:
Difference in flicker-induced vasodilatation of retinal arterioles and venules | Baseline, 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart Center Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Nagele MP, Haider T, Kreysing L, Barthelmes J, Nebunu D, Rossi VA, Hebeisen M, Sudano I, Ruschitzka F, Flammer AJ. Vascular Endothelial Effects of Sacubitril/Valsartan in Heart Failure With Reduced Ejection Fraction: Randomized Controlled Trial. JACC Adv. 2024 Nov 13;3(12):101392. doi: 10.1016/j.jacadv.2024.101392. eCollection 2024 Dec. PMID 39606217